CLINICAL TRIAL: NCT01323452
Title: The Antiviral Efficacy of Entecavir in Chronic Hepatitis B Within the European Network of Excellence (VIRGIL)
Brief Title: Entecavir for Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Prof. Dr. H.L.A. Janssen, Foundation for Liver and Gastrointestinal Research (SLO)
Other Study IDs: VIRGIL
Record Dates: First submitted 2011-03-21; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Entecavir for Chronic Hepatitis B Patients
Keywords: entecavir; hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — entecavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic HBV patients: Patients with chronic hepatitis B Treated for at least 3 months No HIV, HCV or HDV.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — once daily

SUMMARY:
The primary aim of this study is to asses the efficacy (both virological and clinical) and safety of ETV in both NA-naïve and NA-experienced chronic hepatitis B patients, and to explore baseline factors associated with virologic reponse (VR) to ETV.

DETAILED DESCRIPTION:
Chronic hepatitis B is a major health problem, affecting more than 350 million people worldwide. (1) First line treatment consists of pegylated IFN once weekly or oral nucleos(t)ide analogues (NA) once daily. (2) NA target the reverse transcriptase of hepatitis B virus (HBV), and are potent inhibitors of viral replication. In the absence of antiviral drug resistance, continued NA therapy is able to suppress viral replication over prolonged periods, and can prevent clinical progression to liver cirrhosis and hepatocellular carcinoma. (3) Currently approved agents include the nucleoside analogues lamivudine (LAM), telbivudine (LdT), and entecavir (ETV), and the nucleotide analogues adefovir dipivoxil (ADV), and tenofovir disiproxil fumarate (TDF).

Entecavir ETV is a cyclopentyl guanosine analogue, and a potent and selective inhibitor of HBV replication in vitro.(4) In the phase III registration trials it resulted in superior virologic, biochemical and histological efficacy after one year of therapy compared to LAM in both HBeAg-positive and HBeAg-negative chronic HBV patients. (5, 6) Moreover, ETV proved to have a high genetic barrier to resistance with only 1.2% of NA-naïve HBV patients demonstrating genotypic resistance to ETV after five years of ETV monotherapy.(7) In LAM-refractory chronic HBV patients ETV appeared to be less potent and the frequency of resistance was increased. (8, 9) After five years of treatment 51% of LAM-refractory patients showed genotypic ETV resistance, and in 43% a virologic breakthrough was observed as well. (7) Recently we presented the promising results of a large European cohort of patients treated with ETV for a median period of 12 months. We concluded that ETV should not be used in patients with a prior history of LAM-resistance. However, prior treatment with ADV did not influence the efficacy of ETV in these patients.(10)

HBeAg loss or seroconversion In HBeAg positive patients, HBeAg loss or seroconversion is the major objective of NA treatment regimes according to current guidelines. HBeAg loss or seroconversion is usually associated with sustained remission and a very low risk for the development of cirrhosis and hepatocellular carcinoma. (11-13) PEG-IFN induced HBeAg seroconversion was shown to be sustained in 70% after a 3 year follow up. (14) There are some contradictory results concerning NA induced durability of HBeAg loss or seroconversion. First reports on lamuvidine induced HBeAg loss or seroconversion were rather promising.(15-17) However, more recent and also larger studies report much higher relapse rates and predictors of sustainability were proposed. (18-21) The registration trial of entecavir showed a 82% durability after 24 weeks without consolidation therapy.(6) Recently we showed that the durability of HBeAg seroconversion was very poor with 42%, 58% and 74% seroreversion respectively 1,2 and 3 years after seroconversion on different NA treatment regimes. However, only a minority of these patients was treated with the newer and more potent NA. (22)

As the increasing number of patients who experienced treatment failure to different NA treatment regimens poses a growing problem for the clinician, data on the efficacy of ETV in these NA-experienced patient groups is warranted. Furthermore, current guidelines are subject of discussion as durability of NA induced HBeAg loss or seroconversion seems less sustained then expected, and prolonged or maybe infinite therapy may be necessary to prevent long term complications.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for at least 6 months
* Entecavir therapy for at least 3 months

Exclusion Criteria:

* viral co infections
* concomitant antiviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive adult CHB patients treated with ETV monotherapy in 10 large European referral centers
Sampling Method: Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Virological response | 144 weeks after starting Entecavir
  Cumulative probability (%) of patients achieving HBV DNA negativity at week 144

CONTACTS AND LOCATIONS:
Overall Officials: Harry LA Janssen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Mc, Rotterdam, Netherlands